CLINICAL TRIAL: NCT01099644
Title: Phase I Study of Intraperitoneal Radioimmunotherapy With 131I-8H9 for Patients With Desmoplastic Small Round Cell Tumors and Other Solid Tumors Involving the Peritoneum
Brief Title: Intraperitoneal RIT With 131I-8H9 for Pts With DSRCT and Other Solid Tumors Involving the Peritoneum
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Corporate business decision. Not due to safety or efficacy concerns
Sponsor: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-090
Record Dates: First submitted 2010-04-06; First posted 2010-04-07 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Peritoneal Cancer
Keywords: Peritoneum; Desmoplastic Small Round Cell Tumors; Intraperitoneal Radioimmunotherapy; 131 I-8H9; 09-090

ARMS (1):
- 131 I-8H9 (Experimental): This is a phase I study of 131I-8H9 for patients with DSRCT and other 8H9-reactive solid tumors metastatic to the peritoneum.
  Interventions: Biological: 131 I-8H9

INTERVENTIONS:
Biological: 131 I-8H9 — Patients will be administered therapeutic dose of IP 131I-8H9 per the dose escalation regimen. 131I-8H9 pharmacokinetics will be studied by serial blood draws from indwelling venous lines. 131I-8H9 biodistribution will be studied by a single gamma camera scan about 5 days after IP injection where feasible.

SUMMARY:
A phase I study of Intraperitoneal Radioimmunotherapy with 131 I-omburtamab in patients >1 year of age with desmoplastic small round cell tumors and other solid tumors involving the peritoneum.

DETAILED DESCRIPTION:
The purpose of this study is to test the safety of a new medicine called antibody 8H9 injected into the lining of the abdomen or peritoneum, where the tumor is. This medicine is an antibody or protein which binds to certain tumors, including DSCRT. There is a small number of DSCRT which do not bind with 8H9. If the tumor does not bind with 8H9, you might not benefit from this treatment. The investigators want to find out what effects, good and/or bad, it has.

This antibody is made in mice. Radioactive iodine can be bound to this antibody to deliver radiation to the tumor. The investigators wish to determine the safety of radiolabeled 8H9 at different dose levels. This is the first study using 131I-8H9 in the peritoneum.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the diagnosis of (a) DSRCT with peritoneal involvement or (b) other Burtomab-positive solid tumors involving the peritoneum (e.g. adrenocortical carcinoma, Wilm's tumor).
* For tumors other than DSRCT, patients must have a history of tumor progression or recurrence or failure to achieve complete response with standard therapy or <20% chance of long term disease-free survival.
* For tumors other than DSRCT, Burtomab reactivity must be confirmed by immunohistochemistry.
* Patients with DSCRT are not required to have measurable or evaluable disease.
* Patients with tumors other than DSRCT without measurable or evaluable disease will only be considered if they have <20% chance of long term disease-free survival.
* Prior Therapy: At least 4 weeks should have elapsed since any biologic therapy, or immunotherapy. Three weeks should have elapsed since last dose of chemotherapy or radiotherapy.
* Age >1 year and able to cooperate with radiation safety restrictions during therapy period.
* Stem cells: Patients must have an autologous hematopoietic stem cell product cryopreserved and available for re-infusion after 131 I-Burtomab treatment. The minimum dose for hematopoietic stem cells is 2 x 106 CD34+ cells/kg.
* Minimum life expectancy of six weeks as determined by consenting professional.
* Signed informed consent indicating awareness of the investigational nature of this program.

Exclusion Criteria:

* Severe major organ toxicity. Renal, cardiac, hepatic, pulmonary, gastrointestinal and neurologic toxicity should all be grade 1 or less (per NCI CTC version 3 criteria) with the following exceptions: serum AST,ALT and alkaline phosphatase should be ≤5 x upper limit of normal (ULN), serum bilirubin ≤ 3 x ULN and nausea and vomiting should be ≤ grade 2 Patients with myelosuppression are not excluded if ANC ≥ 500/uL.
* Platelet count should be > 50,000/ul and hemoglobin should be > 8gm/dl. Patients may receive platelet or red blood cell transfusions to maintain hemoglobin and platelets at clinical appropriate levels.
* Patients with clinically suspected dense intraperitoneal adhesions preventing adequate IP distribution.
* History of allergy to mouse proteins.
* Patients previously treated with murine monoclonal antibodies will be excluded if they have a HAMA level of >1000U/ml.
* Active serious infections not controlled by antibiotics.
* Pregnant women and women who are breast feeding are excluded for fear of danger to the fetus/infant. Therefore negative pregnancy test is required for all women of child-bearing age, and appropriate contraception is used during the study period. Pregnancy testing will be carried out within two weeks prior to administration of radioiodinated Burtomab in females of childbearing age.
* Inability or unwillingness to comply with radiation safety procedures or protocol requirements.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

PRIMARY OUTCOMES:
Define the toxicity of 131I-8H9 administered intraperitoneally. | weekly
  Assessment of toxicity of 131I-8H9 administered intraperitoneally.

SECONDARY OUTCOMES:
Define maximal tolerated dose (MTD) of 131I-8H9 administered intraperitoneally | 5 years
  Assessment of maximal tolerated dose of 131I-8H9 administered intraperitoneally
Assess pharmacokinetics for 131I-8H9 administered intraperitoneally | 0 hrs, 60 mins, 2 hrs, 8 hrs, 18hrs, 30 hrs, 42hr, 66hrs, 90 hrs, and 114hrs.
  Assessment of the pharmacokinetics for IP 131I-8H9 administered intraperitoneally
Assess response of DSRCT and other solid tumors to 131 I-8H9 administered intraperitoneally | between days 24 and 38
  Assessment of the response of DSRCT and other solid tumors to 131 I-8H9 administered intraperitoneally

CONTACTS AND LOCATIONS:
Overall Officials: Shakeel Modak, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Modak S, Zanzonico P, Grkovski M, Slotkin EK, Carrasquillo JA, Lyashchenko SK, Lewis JS, Cheung IY, Heaton T, LaQuaglia MP, Cheung NV, Pandit-Taskar N. B7H3-Directed Intraperitoneal Radioimmunotherapy With Radioiodinated Omburtamab for Desmoplastic Small Round Cell Tumor and Other Peritoneal Tumors: Results of a Phase I Study. J Clin Oncol. 2020 Dec 20;38(36):4283-4291. doi: 10.1200/JCO.20.01974. Epub 2020 Oct 29. PMID 33119478
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org